CLINICAL TRIAL: NCT01801670
Title: A Phase IV Study Of The Impact Of Vorinostat On Cellular Signaling And Cytokine Production In Cutaneous T-Cell Lymphoma Patients With Pruritus
Brief Title: Impact of Vorinostat on Pruritus Signaling Pathways - Merck Study
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment was too slow, so no participants were ever enrolled.
Sponsor: Boston University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 30121
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Pruritus
Keywords: itch; pruritus; skin; vorinostat; cutaneous T-cell lymphoma; mycosis fungoides
MeSH Terms: conditions — Pruritus; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples Skin biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MF patients for blood & biopsy: Participants who are cared for at Boston Medical Center will first be assessed by physicians of the CTCL multi-specialty clinic if vorinostat, administered per standard of care, is an appropriate therapy for their CTCL. The decision to invite patients to participate in this study is (1) separate from the above described clinical decision to utilize vorinostat, and (2) will be offered subsequent to the clinical decision to utilize vorinostat. Vorinostat (Zolinza) will be administered as follows: each subject will receive each month for the first 3 months (cycle 1 to 3) 3 capsules of vorinostat 100 mg po daily. For months 4-6 (cycles 4 to 6), subjects will receive each month for 4 capsules of vorinostat 100 mg po daily.
  Interventions: Procedure: Biopsy; Procedure: Blood

INTERVENTIONS:
Procedure: Biopsy — Two 6 mm skin punch biopsies (one from pruritic skin and from involved non pruritic skin).
Procedure: Blood — Peripheral blood (10 mls) to be drawn and used for cytokine analysis.

SUMMARY:
Mycosis Fungoides (MF) is a rare malignancy in the United States. It is the most common form of cutaneous T-cell lymphoma (CTCL). Sézary syndrome (SS) is the most severe and leukemic form of CTCL. Pruritus, or itch, is defined as an unpleasant sensation that elicits the desire to scratch. Severe itch is a manifestation of all forms of MF, especially those with patch/plaque and folliculotropic variants, as well as in Sezary patients. While severe itch causes great suffering for patients, the pathogenesis of itch in MF and Sezary syndrome is complex and not well understood. It is thought that various chemical mediators are produced by the malignant cells to cause itch. Vorinostat, an FDA approved therapy for the treatment of MF, has also been reported to relieve pruritis. The goal of the study is to evaluate how vorinostat affects different chemicals in the skin that have been known to cause itch. This is a single center, non-randomized study designed to obtain and test blood and skin tissue samples take at various time-points over 6 months in patients who are prescribed vorinostat per standard of care treatment. Samples from pruritic and non-pruritic skin and blood of MF and Sezary patients will be evaluated for the presence of chemicals thought to be important in the cause of itch in these diseases. This evaluation will include immunohistochemistry, RT-PCR, and ELISA assays. The results from this study may help define how vorinostat decreases itch in patients with MF and Sezary Syndrome.

DETAILED DESCRIPTION:
Mycosis Fungoides (MF) is a rare malignancy in the United States. It is the most common form of cutaneous T-cell lymphoma (CTCL). Sézary syndrome (SS) is the most severe and leukemic form of CTCL. Severe pruritus is a manifestation of the SS and also affects patients with MF. Severe pruritus is a manifestation of SS and also a common symptom among patients with MF. Pruritus can significantly impact on quality of life. In one national survey of the impact of MF on patients' health-related quality of life (HRQOL), the majority of survey respondents (88%) reported being bothered by pruritus.

The pathogenesis of pruritus is complex and not well understood. It affects a majority of patients with mycosis fungoides (MF) and is most severe in Sézary syndrome (SS), the leukemic form of cutaneous T-cell lymphoma. Chemical or physical stimuli that perturb, without damaging, only the epidermis (the outer most layer of the skin), elicit the symptom of pruritus. The perception of itch is abolished if the epidermis is removed. This observation and the data on PAR2 expression on nerve fibers indicate that pruritus in inflammatory skin disorders including MF/SS is likely to have a neuroepidermal origin or be mediated by molecules that percolate to the epidermis from inflammatory cells in the dermis. In this regard, MF/SS are characterized histologically by infiltration of the epidermis by neoplastic T cells (epidermotropism), and in some of these cases, the neoplastic cells form collections of 2-3 cells around epidermal Langerhans cells (Pautrier microabscess). Neoplastic cells of advanced MF/SS typically are polarized to secrete TH2 cytokines. It has been hypothesized that the accumulation of neoplastic cells in skin lesions promotes a shift from a TH1 predominant cytokine profile in early MF to a TH2 predominant cytokine profile in advanced disease 4. The shift to TH2 production coincides with impaired immune responses, eosinophilia, and high levels of IgE in the blood. Severe pruritus is more frequent in patients with advanced MF/SS suggesting that tumor burden or cytokines elaborated by activated tumor cells may be correlated to intensity of pruritus.

While it is not clear which cells contributed to the TH2 cytokine shift, studies of T-cells isolated from skin and blood of affected patients showed activation of the signaling molecule, STAT3. In CTCL lines, constitutively activated STAT3 mediates IL-5 production (principal regulator of eosinophilia) and IL-13 (favors antibody responses) 5. Moreover, IL-31 also seems to signal through STAT3 in one lung model. Current treatments of pruritus are aimed towards symptomatic relief although these do not address the mechanism of pruritus. If neoplastic cells are producing IL-31 or other pruritogenic factor as we propose, then any treatment that eliminates these cells will also be effective for pruritus. To date, effectively improving pruritus and the disease manifestations is not always possible especially in advanced MF or SS.

Vorinostat is a FDA approved histone deacetylase inhibitor for the treatment of the cutaneous manifestations of patients with cutaneous T-cell lymphoma (MF/SS) who have progressive, persistent, or recurrent disease on or following 2 systemic therapies. Vorinostat induces differentiation, growth arrest, and/or apoptosis of malignant cells both in vitro and in vivo and has shown clinical responses in approximately 30% of patients with advanced MF/SS 7. Overall, 32% of patients with severe pruritus had relief of this symptom, and it was observed that the relief of pruritus often presaged the clinical response, especially in SS. This suggests to us that the gene modulating effects of vorinostat might be directly inhibiting expression of IL-31 or other cytokines that mediate pruritus in MF/SS. IL-31 appears to be implicated in pruritus of atopic dermatitis. 8 Recently, studies have demonstrated that itch can be mediated by a novel cysteine protease and that proteinase-activated receptor-2 plays an important role in itch signaling pathways. 9, 10 In another recent study, substance P has been implicated in itch pathophysiology. In one small case series of patients with CTCL, the efficacy of aprepitant was evaluated11. Aprepitant is a substance P antagonist that blocks the neurokinin 1 (NK1) receptor. Substance P has a role in the physiology of unmyelinated C-fibers in the skin that convey both pain and pruritus and has the ability to modulate mast cell functioning.

Data from skin biopsies have shown that successful treatment with vorinostat is associated with decreased dermal and epidermal lymphocytes, a shift from nuclear to cytoplasmic p-STAT-3 staining, and decreased CD31-positive dermal vessels. This was not confirmed in another study. Vorinostat has been postulated to indirectly inactivate STAT proteins that drive cellular proliferation and TH2 cytokine expression. Researchers observed that in skin biopsies of patients enrolled in the vorinostat stage IIB trial, nuclear accumulation of STAT1 and high levels of nuclear pSTAT3 in malignant T cells correlated with a lack of clinical response. To date, there has been no evaluation of STAT3 proteins and TH2 cytokines in pruritic versus non-pruritic skin lesions of CTCL. Signal transducers and activators of transcription (STATS) are important to active transcription of cellular proteins including cytokines. Constitutive activation of STATs has been shown to be a feature of MF/SS.

Study Rationale:

Since pruritus is a common manifestation of the disease that significantly impacts on patient's quality of life and that oral vorinostat provides clinical relief from pruritus in treated patients, understanding the mechanisms of action of vorinostat on cytokines implicated in pruritus will shed light on its therapeutic effect. In particular, because we believe that a reduction in pSTAT3 activity as evidenced by fewer and/or less strongly stained tumor cells may be taking place in patients responding to therapy and reporting decrease pruritus. Thus, understanding the extent of STAT3 protein aberration and cytokine expression (IL-31) in pruritic skin lesions could significantly contribute to our understanding of the mechanism of pruritus in MF/SS and to how vorinostat relieves this serious symptom.

Objectives/Hypothesis It is hypothesized that skin tissue expression of pSTAT3, IL-31, and cathepsin S will correlate with response to vorinostat, a recently FDA approved therapy for MF and SS, decreasing in expression with relief of pruritus.

Methods: Dosing and Frequency of Drug

Participants who are cared for at Boston Medical Center will first be assessed by physicians of the CTCL multi-specialty clinic if vorinostat, administered per standard of care, is an appropriate therapy for their CTCL. The decision to invite patients to participate in this study is (1) separate from the above described clinical decision to utilize vorinostat, and (2) will be offered subsequent to the clinical decision to utilize vorinostat. There is no placebo group for this study. Up to ten participants are desired for this study.

Three biopsies will be taken: (1) at baseline; (2) after 4 weeks of 300 mg daily vorinostat, and (3) if tolerated, after 4 more weeks of 400 mg daily vorinostat. At each time point, up to 2 biopsies will be taken depending on if 1 or both skin types are present (itchy vs non-itchy) at that time point and whether or not itchy or non-itchy skin shows a lesion. For each time point and each skin type, pSTAT3 staining will be measured as strong (2+), weak (1+), none (0). At each time point, patients will report the extent of their pruritus on a visual analogue score (VAS) from 0-100 mm (0, no pruritus; 100, worst imaginable pruritus). Meaningful change in pruritus will be a change in VAS score of 30 mm or more from baseline to the third time point (a change measure that will also be computed for all endpoints; the baseline to time 3 measure being of primary clinical interest).

Sample Size/Accrual Rate: The total enrollment planned is 10 patients at a rate of 1-2 patients per month. With 10 subjects, for our primary hypothesis (correlation of staining intensity with self-reported degree of pruritis) we can detect a Spearman rank correlation coefficient as small as 0.75 for a one-sided test with 80% power (a directional hypothesis that is reasonable) or one as small as 0.80 for a two-sided hypothesis. In each case, these coefficients are of clear clinical relevance and are plausible given the nature of the measures. For the hypothesis of equal changes between treated and control areas on the same individuals, we propose using paired data analyses such as paired t-tests and Wilcoxon rank sum tests. For a sample size of 10 and 80% power, a paired t-test can detect an effect size of 0.996 or greater for a two-sided test and an effect size of 0.853 or greater for a one-sided test. These effect sizes are large but are within reason to expect for a clinically effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients w/ histologically confirmed mycosis fungoides stage IB to IVA eligible to receive oral vorinostat
* Patients w/ stage IB to IV reporting pruritus
* Patients age 18-85 years, of any race, sex, and ethnicity
* Life expectancy > 24 weeks
* Patient must have performance status of ≤2 on the ECOG Performance Scale
* Patients w/ a min. of 3 weeks since their last systemic treatment
* Women who are not pregnant, lactating, or of childbearing potential
* Female patients w/ reproductive potential must use an adequate contraceptive method during treatment and for three months after completing treatment
* Male patient w/ reproductive potential, agrees to use an adequate method of contraception for the duration of the study and for 30 days beyond the duration of study
* Patients, or legal representative must to be willing to adhere to the protocol, and sign an Informed Patient Consent Form prior to entry into the study
* Patients must not be on any other investigational device/drug treatment for MF/SS
* Patient is available for periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study
* Eligibility of patients receiving medications or substances known or with the potential to affect the activity or pharmacokinetics of vorinostat will be determined by the Principal Investigator
* Patient must have adequate organ function as indicated by laboratory values

Exclusion Criteria:

* Patients w/ a recent cardiac history, such as a myocardial infarct within the last year, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Patients w/ a history of liver damage (2.5 x normal ALT, AST), leukopenia, or thrombocytopenia
* Women who are pregnant or nursing a child
* Patients w/ severe emotional, behavioral or psychiatric problems that, in the opinion of the investigator, would result in poor compliance with the treatment regimen
* Patients who have received and histone deacetylase inhibitor within the last 6 months
* Patients receiving valproic acid will be excluded unless there has been a wash-out period of 30 or more days
* Patients who will have received systemic therapy, radiation therapy or phototherapy within 3 weeks prior to initial dosing with study drugs or who has not recovered from adverse events due to agents administered more than 3 weeks earlier
* QTc prolongation greater than 500ms
* Patient w/ a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled
* Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years or are considered by their physician to be at less than 30% risk of relapse
* Patient is on any systemic steroids that have not been stabilized during the 3 weeks prior to the start of the study drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patient is, at the time of signing informed consent, a regular user of any illicit drugs, substance abuse or had a recent history (within last year) of drug or alcohol abuse
* Patient has uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including, but not limited to: active infection, acute or chronic graft versus host disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric conditions
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate
* HIV-positive patients will be ineligible
* Patients w/ known history of Hepatitis B or C are excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with CTCL-mycosis fungoides type treated at Boston Medical Center and that have, independent of this study, already agreed to start vorinostat according to the stand-of-care guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
the percentage change in pSTAT3 expression among patients reporting a relief in their pruritus, irrespective of lesion clearing | 6 months
  For each time point and each skin type, pSTAT3 staining will be measured as strong (2+), weak (1+), none (0). At each time point, patients will report pruritus on a visual analogue score (VAS) from 0-100 mm (0, none; 100, worst imaginable). Meaningful change in pruritus is a change in VAS score of 30 mm or more from baseline to the third time point (a change measure that will also be computed for all endpoints; the baseline to time 3 measure being of primary clinical interest).
  Spearman rank correlation will examine the significance of the association between the change in cytoplasmic staining intensity and change in pruritus as assessed by subjects with the visual analog scale, neither of which will be assumed to follow a Gaussian distribution.
  For descriptive purposes only, analyses will also be performed stratified on pruritis stage at baseline (early stage I-IIA vs. late stage IIB-IVB and pruritus, mild VAS less than 40 vs. moderate to severe VAS greater than 40, up to 100).

SECONDARY OUTCOMES:
IL-31 amount and intensity of cathepsin S expression | 6 months
  IL31 amount and cathepsin S intensity of expression will be determined at 3 time points described above and also from itchy and non-itchy skin at each time point. The goal is to determine if there is an association between a change (presumably a decrease) in these targets and an improvement in pruritus as reported by the VAS score.
  Spearman rank correlation will examine the significance of the association between the change in amount of IL-31 or level of cathepsin S expression and change in pruritus as assessed by subjects with the visual analog scale, neither of which will be assumed to follow a Gaussian distribution.
  For this data, taken in separate locations (treatment, control) on the same individuals, we will perform paired t-tests or non-parametric Wilcoxon signed rank tests as appropriate.
percentage of vasodilatory peptidergic nerves at the dermoepidermal junction as a percentage of total nerves | 6 months
  The total nerve length of all nerves and the total nerve length of nerves expressing vasodilatory peptidergic markers will be determined in the skin biopsies at 3 time points described above, and the percentage calculated.
  Spearman rank correlation will examine the significance of the association between the change in the above percentage of nerves and change in pruritus as assessed by subjects with the visual analog scale, neither of which will be assumed to follow a Gaussian distribution.
  For this data taken in separate locations (treatment, control) on the same individuals, we will perform paired t-tests or non-parametric Wilcoxon signed rank tests as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Deon Wolpowitz, MD, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States